CLINICAL TRIAL: NCT04995666
Title: Hearing Aid Quality Check and Reliability Study
Brief Title: Hearing Aid Quality and Reliability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-368
Record Dates: First submitted 2021-06-11; First posted 2021-08-09 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hearing Aid (Experimental): Participants will wear Phonak rechargeable Audeo hearing aids
  Interventions: Device: Phonak Audeo hearing aid

INTERVENTIONS:
Device: Phonak Audeo hearing aid — Rechargeable hearing aid

SUMMARY:
Quality and reliability study of hearing aid. Adults with mild to severe hearing loss will wear hearing aids daily for approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with mild to moderate severe sensorineural hearing loss
* Adults who were able to incorporate some type of physical activity into their day (i.e walking, excercise, gardening, etc.)

Exclusion Criteria:

* Unable or unwilling to wear study devices during a home trial
* Unable or unwilling to come to lab for study visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hearing Aid
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hearing Aid
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 70 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Electroacoustic Evaluation of Hearing Aids in Accordance With Manufacturer Specifications, Day 1
Description: Test box electroacoustic measurements of hearing aid done at full on settings must meet manufacturer product specifications per manufacturer data sheet. This includes maximum and high frequency average output sound pressure level, maximum and high frequency average acoustic gain, frequency response range, total harmonic distortion and equivalent input noise level. This is done using an Audioscan Verifit2 electroacoustic analyzer.
  Electroacoustic measurements listed above will also be taken with hearing aid set to user settings, as a baseline measure for all future appointments.
Time Frame: Day 1 of study
Population: All devices dispensed to study participants on day 1 of study tested on electroacoustic verification equipment
Measure: Count of Units; unit: hearing aid devices
Units Other Than Participants: hearing aid devices
Arm/Group | Hearing Aid
Number analyzed (Participants) | 19
Number analyzed (hearing aid devices) | 38
hearing aid devices
  Number of units that PASS manufacturer specifications | 38
  Number of units that FAIL manufacturer specifications | 0

2. Primary Outcome: Electroacoustic Evaluation of Hearing Aids in Accordance With Manufacturer Specifications, Day 45
Description: Test box electroacoustic measurements (using the Audioscan Verifit 2 Electroacoustic Analyzer) of hearing aid done at user gain settings after daily use for extended period of time. Results will be compared to baseline electroacoustic measures taken on day 1 of study. A "pass" means that devices were within tolerance levels (per ANSI S3.22-2014) of baseline measures. A "fail" means that devices were not within tolerance levels of one or more baseline measures (i.e. output, gain, frequency range, total harmonic distortion, or equivalent input noise level).
Time Frame: Day 45 of study
Population: All devices dispensed to study participants on day 1 of study tested on electroacoustic verification equipment
Measure: Count of Units; unit: hearing aid devices
Units Other Than Participants: hearing aid devices
Arm/Group | Hearing Aid
Number analyzed (Participants) | 19
Number analyzed (hearing aid devices) | 38
hearing aid devices
  Number of devices that PASS manufacturer specifications specifications | 38
  Number of devices that FAIL manufacturer specifications | 0

3. Primary Outcome: Electroacoustic Evaluation of Hearing Aids in Accordance With Manufacturer Specifications, Day 90
Description: Test box electroacoustic measurements of hearing aid done at user gain settings after daily use for extended period of time. Test box electroacoustic measurements of hearing aid done at user gain settings after daily use for extended period of time. Results will be compared to baseline electroacoustic measures taken on day 1 of study. A "pass" means that devices were within tolerance levels (per ANSI S3.22-2014) of baseline measures. A "fail" means that devices were not within tolerance levels of one or more baseline measures (i.e. output, gain, frequency range, total harmonic distortion, or equivalent input noise level).
Time Frame: Day 90 of study
Population: All devices dispensed to study participants on day 1 of study tested on electroacoustic verification equipment. One participant lost a device, therefore total number of devices analyzed on Day 90 is 37.
Measure: Count of Units; unit: hearing aid devices
Units Other Than Participants: hearing aid devices
Arm/Group | Hearing Aid
Number analyzed (Participants) | 19
Number analyzed (hearing aid devices) | 37
hearing aid devices
  Number of devices that PASS manufacturer specifications | 35
  Number of devices that FAIL manufacturer specifications | 2

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Hearing Aid
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hearing Aid (N=19)
Complication (Ear and labyrinth disorders) | 1 (1) — Participant reported pain and moisture in left ear 3 weeks after hearing aid fitting. Issue resolved after seeing physician and receiving medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04995666/Prot_SAP_000.pdf